CLINICAL TRIAL: NCT04236882
Title: A Randomized-Crossover Sleep and Physical Activity (PA) Intervention for Overweight/Obese and Sedentary African Americans
Brief Title: Sleep and Physical Activity Intervention for Increasing Physical Activity in Overweight or Obese and Sedentary African Americans
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0568; NCI-2019-07036 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0568 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-04; First posted 2020-01-22 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Behavioral Disorder; Endocrine System Disorder
MeSH Terms: conditions — Mental Disorders; Endocrine System Diseases | interventions — Focus Groups; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Focus group and interview (focus group, interview) (Experimental): Participants attend either a focus group or interview about the sleep intervention and sleep-related problems over 90 minutes.
  Interventions: Other: Focus Group; Other: Interview; Other: Questionnaire Administration
- Group I (sleep intervention, health coaching session) (Experimental): Participants receive a web-based sleep intervention weekly during weeks 1-4. Participants then receive 2 web-based health coaching sessions over 30-45 minutes consisting of topics such as healthy shopping, increasing physical activity, identifying barriers, and eating out during weeks 5-9. Participants may optionally complete an interview over 1 hour at week 9.
  Interventions: Other: Internet-Based Intervention; Other: Interview; Other: Questionnaire Administration
- Group II (health coaching session, sleep intervention) (Experimental): Participants receive 2 web-based health coaching sessions over 30-45 minutes consisting of topics such as healthy shopping, increasing physical activity, identifying barriers, and eating out during weeks 1-4. Participants then receive a web-based sleep intervention weekly during weeks 5-9. Participants may optionally complete an interview over 1 hour at week 9.
  Interventions: Other: Internet-Based Intervention; Other: Interview; Other: Questionnaire Administration
- Group III (health education material, counseling session) (Active Comparator): Participants receive educational material on healthy homes. Participants also receive 2 web-based counseling sessions over 30-45 minutes consisting of topics such as indoor air quality, CPR and first aid, and emergency preparedness at weeks 1 and 3. Participants may optionally complete an interview over 1 hour at week 9.
  Interventions: Behavioral: Health Education; Other: Internet-Based Intervention; Other: Interview; Other: Questionnaire Administration

INTERVENTIONS:
Other: Focus Group — Attend focus group
  Arms: Focus group and interview (focus group, interview)
Behavioral: Health Education — Receive educational material on healthy homes
  Arms: Group III (health education material, counseling session)
Other: Internet-Based Intervention — Receive web-based sleep intervention
  Arms: Group I (sleep intervention, health coaching session); Group II (health coaching session, sleep intervention)
Other: Internet-Based Intervention — Receive web-based health coaching sessions
  Arms: Group I (sleep intervention, health coaching session); Group II (health coaching session, sleep intervention)
Other: Internet-Based Intervention — Receive web-based counseling sessions
  Arms: Group III (health education material, counseling session)
Other: Interview — Complete interview
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well sleep and physical activity interventions work in increasing the physical activity of overweight or obese and sedentary African Americans. Sleep and physical activity interventions may help to increase physical activity among overweight and obese African American adults who do not get enough exercise.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility and satisfaction of a brief sleep intervention prior to or following a physical activity (PA) intervention and a contact control among overweight/obese sedentary African Americans.

II. Examine experiences of sleep among overweight/obese sedentary African Americans using qualitative focus groups/individual interviews.

SECONDARY OBJECTIVES:

I. Pilot test and evaluate the efficacy and sequential effects of a brief sleep intervention prior to or following a PA intervention in improving sleep, increasing physical activity, and reducing sedentary behavior, compared to a contact control group.

II. Explore the correlations among psychosocial (e.g., perceived stress, affect, neighborhood characteristics), biomarker (e.g., non-fasting glucose levels, blood pressure), and health behavior (e.g., diet and sedentary behavior) with sleep and PA.

OUTLINE:

FOCUS GROUPS AND INTERVIEWS: Participants attend either a focus group or interview about the sleep intervention and sleep-related problems over 90 minutes.

Participants are randomized to 1 of 3 groups.

GROUP I: Participants receive a web-based sleep intervention weekly during weeks 1-4. Participants then receive 2 web-based health coaching sessions over 30-45 minutes consisting of topics such as healthy shopping, increasing physical activity, identifying barriers, and eating out during weeks 5-9. Participants may optionally complete an interview over 1 hour at week 9.

GROUP II: Participants receive 2 web-based health coaching sessions over 30-45 minutes consisting of topics such as healthy shopping, increasing physical activity, identifying barriers, and eating out during weeks 1-4. Participants then receive a web-based sleep intervention weekly during weeks 5-9. Participants may optionally complete an interview over 1 hour at week 9.

GROUP III: Participants receive educational material on healthy homes. Participants also receive 2 web-based counseling sessions over 30-45 minutes consisting of topics such as indoor air quality, cardiopulmonary resuscitation (CPR) and first aid, and emergency preparedness at weeks 1 and 3. Participants may optionally complete an interview over 1 hour at week 9.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (not meeting Physical Activity Guidelines)
* Overweight and/or obese adults (body mass index range: 25.0 or greater)
* Average habitual sleep duration of =< 6 hours
* Access to internet
* Self-identify as black or African American
* Able to engage in moderate intensity physical activity as determined by the Physical Activity Readiness Questionnaire (PAR-Q) or by physicians clearance (letter from physician or nurse practitioner) if endorsing any items on the PAR-Q

Exclusion Criteria:

* Pre-existing sleep disorder (i.e., insomnia, sleep apnea, restless leg syndrome, narcolepsy, and sleep walking disorder via self-report)
* High risk for obstructive sleep apnea (i.e., STOP-BANG score > 5)
* Psychiatric disorder (current risk of severe depression as measured by Center for Epidemiologic Studies Depression Scale [CESD] > 15 with/without past history of diagnosed Diagnostic and Statistical Manual of Mental Disorders [DSM-V] disorder)
* Self-reported physician diagnosed thyroid condition that is not currently being treated
* Shift work or employment that requires weekly flights to a different time zone or overnight travel
* Enrolled in weight management program
* Excessive caffeine intake (> 400 mg caffeine intake/day or the equivalent of > 4 cups of coffee)
* Plans to change residence out of Houston within the next 3 months
* Self-reported pregnancy or less than 4 months postpartum
* Participated in formative focus groups/individual interviews for this study
* Blood pressure readings >= 140/90 mm or by physicians clearance (letter from physician or nurse practitioner) if blood pressure reading >= 140/90 mm Hg
* Another household member is enrolled in the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-10-04 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Determine the f easibility of a brief sleep intervention prior to or following a physical activity (PA) intervention | Up to 9 weeks
Satisfaction of a brief sleep intervention prior to or following a PA intervention | Up to 9 weeks
Sleep experiences | Up to 9 weeks
  Will examine experiences of sleep among overweight/obese sedentary African Americans using qualitative focus groups.

SECONDARY OUTCOMES:
Sleep improvement | At 9 weeks
  Will pilot test and evaluate the efficacy of a brief sleep intervention prior to or following a PA intervention in improving sleep.
Physical activity increase | At 9 weeks
  Will pilot test and evaluate the efficacy of a brief sleep intervention prior to or following a PA intervention in increasing physical activity.
Sedentary behavior reduction | At 9 weeks
  Will pilot test and evaluate the efficacy of a brief sleep intervention prior to or following a PA intervention in reducing sedentary behavior.

OTHER OUTCOMES:
Psychosocial behavior | Up to 9 weeks
  Will explore the correlations among psychosocial behavior (e.g., perceived stress, affect, neighborhood characteristics) with sleep and PA.
Biomarker analysis | Up to 9 weeks
  Will explore the correlations among biomarker levels (e.g., non-fasting glucose levels, blood pressure) with sleep and PA.
Health behavior | Up to 9 weeks
  Will explore the correlations among health behavior (e.g., diet and sedentary behavior) with sleep and PA.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna McNeill, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - The Univeristy of Texas M. D. Anderson Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org